CLINICAL TRIAL: NCT03408093
Title: Cross-sectional Retrospective Study of Therapeutic Compliance in Patients With Multiple Sclerosis Treated With Interferon Beta-1b
Brief Title: Study of Betaferon Adherence in Patients With Multiple Sclerosis Treated With Interferon Beta-1b
Acronym: ADHERENCE
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 2008/01880
Record Dates: First submitted 2018-01-08; First posted 2018-01-23 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Multiple Sclerosis
Keywords: Interferon beta-1b (INFb-1b); Multiple Sclerosis (MS); Relapsing-remitting MS (RRMS); Secondary progressive MS (SPMS); Clinically isolated syndrome (CIS)
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Interferon beta-1b: Patients with CIS, RRMS or SPMS who had more than 6 months in treatment
  Interventions: Drug: Interferon beta-1b (Betaseron, BAY86-5046)

INTERVENTIONS:
Drug: Interferon beta-1b (Betaseron, BAY86-5046) — Interferon beta-1b (INFb-1b) was used at the standard dose of 250 mg/ml.

SUMMARY:
The primary objective of the study is to evaluate the adherence to the treatment with interferon beta-1b, in patients diagnosed with isolated syndrome (CIS), relapsing-remitting multiple sclerosis (RRMS), or secondary progressive multiple sclerosis (SPMS) who had more than 6 months in treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsing-remitting MS (RRMS), secondary progressive MS (SPMS) or patients with a first outbreak or clinically isolated syndrome (CIS) that carry more than 6 months in treatment with interferon beta-1b

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included patients who had been on interferon beta-1b for more than 6 months and who agreed to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2009-02-03 (Actual); Primary Completion 2010-03-30 (Actual); Study Completion 2010-03-30 (Actual)

PRIMARY OUTCOMES:
Self-reported adherence to INFb-1b in the previous four weeks assessed by Morisky-Green (MG) test | Four weeks just before baseline visit

SECONDARY OUTCOMES:
Demographic data | At baseline
  Age, sex, marital status, education level, employment status
Number of patients with MS diagnosis | At baseline
Age at first episode and at diagnosis | At baseline
Time since last relapse | At baseline
Assessment of general health status using data from a questionnaire or from their clinical history collected by the investigator team | At baseline
Expanded Disability Status Scale (EDSS) to assess the degree of disability caused by MS | At baseline
  The EDSS quantifies the disability in eight functional systems (FS) and allows neurologists to assign a level of Functional System in each of them caused by multiple sclerosis.
Number of patients with adverse events during the last month | Four weeks just before baseline visit
Clinical setting characteristics like existence of MS unit | At baseline
  The existence of Multiple Sclerosis Unit was evaluated bearing in mind if the hospital had or had not available a Multiple Sclerosis Unit into the hospital Neurology Department.
Time on INFb-1b therapy | At baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer

REFERENCES:
- [Result] Fernandez O, Aguera E, Izquierdo G, Millan-Pascual J, Ramio I Torrenta L, Oliva P, Argente J, Berdei Y, Soler JM, Carmona O, Errea JM, Farres J; Group on Adherence to IFNb-1b in Spain. Adherence to interferon beta-1b treatment in patients with multiple sclerosis in Spain. PLoS One. 2012;7(5):e35600. doi: 10.1371/journal.pone.0035600. Epub 2012 May 16. PMID 22615737